CLINICAL TRIAL: NCT07348263
Title: International Multicentre Cohort Study on Clinical Manifestations and Response to Therapy in Juvenile Onset Eosinophilic Fasciitis
Brief Title: EFESO: Study on Juvenile Onset Eosinophilic Fasciitis
Status: Recruiting | Type: Observational
Sponsor: Meyer Children's Hospital IRCCS (Other)
Responsible Party: Principal Investigator, Gabriele Simonini, MD, Meyer Children's Hospital IRCCS
Other Study IDs: EFESO
Record Dates: First submitted 2026-01-09; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Eosinophilic Fasciitis
Keywords: Eosinophilic Fasciitis; Juvenile eosinophilic fasciitis; juvenile scleroderma; sclerosing disorders
MeSH Terms: conditions — Eosinophilic Fasciitis; Juvenile-onset scleroderma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Juvenile eosinophilic fasciitis: Age < 18 years at diagnosis
  - The study will include two different populations:
  1. Patients who have received a diagnosis of JEF based on deep fascial biopsy characteristics.
  2. Patients who have received a diagnosis of JEF based on typical MRI findings, but without performing a deep fascial biopsy.

SUMMARY:
Eosinophilic fasciitis is a connective tissue disorder characterized by inflammation of the muscle fasciae, which is very rare in children. In juvenile-onset eosinophilic fasciitis (JEF), there may be severe joint involvement and skin manifestations may be less prevalent than in adults. It represents an important differential diagnosis of both juvenile-onset systemic sclerosis and localized scleroderma, and the correct classification of these patients is necessary to define a targeted diagnostic-therapeutic pathway. The diagnostic criteria proposed for eosinophilic fasciitis in the adult population (Pinal-Fernandez et al. 20145; JInnin M 20186) do not necessarily require confirmation by skin biopsy, currently the "gold standard," which is an invasive procedure for pediatric patients; however, these criteria have never been directly applied to the pediatric population. From a therapeutic point of view, the combination of glucocorticoids and methotrexate is recommended for both adults and pediatric patients, but the data supporting this treatment in children are very limited, and there are no studies comparing the therapeutic approaches currently in use in pediatrics. Finally, there are no studies in the literature documenting the long-term prognosis of these patients in terms of functional limitations, quality of life, or complications related to the disease or treatments.

ELIGIBILITY:
Inclusion criterai:

All patients diagnosed from 2000 to 31/12/2026

* minimum follow-up 6 months
* Age <18 years at diagnosis;
* All patients whose informed consent is collected in accordance with current local legislation will also be considered enrollable.

Exclusion Criteria:

* Age ≥18 years at diagnosis;
* Unwilling to participate into the study;
* A follow-up period < 6 months.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study will include patients diagnosed with eosinophilic fasciitis before <18 years of age, separated into two different populations:
  Patients who received a diagnosis of JEF based on deep fascial biopsy features. Patients who received a diagnosis of JEF based on typical MRI findings but without deep fascial biopsy.
  Patients with localized or systemic scleroderma who underwent deep fascial biopsy, in a 1:1 ratio with patients with juvenile eosinophilic fasciitis will be enrolled as a comparison group
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2027-05-15 (Estimated)

PRIMARY OUTCOMES:
Clinical and laboratory features | 2025-2027
  Describe the clinical and laboratory features at presentation and during follow-up, including the extent of skin involvement and extracutaneous manifestations, of patients diagnosed with JEF.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (2):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - SUNY Upstate Pediatric Rheumatology, Syracuse, New York
- Children's Hospital Zagreb, Zagreb, Croatia
- Meyer Children's Hospital IRCCS, Florence, FI, Italy
- Iuliu Hatieganu University of Medicine and Pharmacy, Cluj-Napoca, Romania
- Astrid Lindgren Children's Hospital, Solna, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided